CLINICAL TRIAL: NCT00003268
Title: A Phase I Study of Cytosine Arabinoside, Idarubicin, and Amifostine as Induction Therapy for Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Amifostine and Combination Chemotherapy in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: TJUH-980407; CDR0000066164 (Registry Identifier: PDQ (Physician Data Query)); ALZA-97-040-ii; NCI-V98-1395
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2003-10

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute monoblastic leukemia and acute monocytic leukemia (M5); adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute megakaryoblastic leukemia (M7); drug/agent toxicity by tissue/organ; adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Leukemia; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Amifostine; Cytarabine; Idarubicin

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cytarabine
Drug: idarubicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of amifostine in treating patients with newly diagnosed acute myeloid leukemia who are receiving idarubicin plus cytarabine.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether amifostine provides systemic protection against the nonhematologic side effects of idarubicin (IDR) during induction therapy of acute myeloid leukemia (AML), allowing the dose of idarubicin to be escalated.
* Determine the maximum tolerated dose of idarubicin when amifostine is used as a chemotherapy protectant.
* Determine the incidence and severity of dose limiting hypotension in patients receiving amifostine and the ability to offset this side effect with vasoconstrictive agents.
* Determine whether any additional side effects of amifostine are dose limiting in patients with AML treated with IDR and cytarabine (ARA-C).
* Monitor the frequency of alopecia, mucositis, diarrhea, and septicemia involving enteric pathogens in these patients.
* Determine the requirement for intravenous hyperalimentation in patients receiving amifostine, IDR, and ARA-C.

OUTLINE: This is a dose escalation study of idarubicin (IDR).

Patients receive amifostine IV over 15 minutes, followed 15-30 minutes later by chemotherapy. Idarubicin IV is administered over 15 minutes on days 1-3. Cytarabine is administered by continuous infusion on days 1-7. Patients may receive 1 additional course of treatment, if necessary.

Cohorts of 3-6 patients each are treated at each dose level of idarubicin. Dose escalation is discontinued when 2 or more patients experience dose limiting toxicity.

Patients are followed at 3 months.

PROJECTED ACCRUAL: A maximum of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute myeloid leukemia (AML)

  * M0-M2, M4-M7
  * Histologically proven by bone marrow aspirate and biopsy (requirement may be waived for patients with overt leukemia in the peripheral blood)
  * M3 (acute promyelocytic leukemia) patients excluded unless already treated with trans retinoic acid
* Evaluable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%
* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Not specified

Hepatic:

* SGOT/SGPT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* Ejection fraction at least 50%
* Must be able to stop taking antihypertensive medication 24 hours prior to cytarabine administration

Other:

* No preexisting severe organ dysfunction
* No history of underlying medical or psychiatric illness that may impair the patient's ability to participate in the study
* Not pregnant or nursing
* Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior cytotoxic therapy for AML
* No prior amifostine
* At least 1 month since chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 1 month since radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-01; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Flomenberg, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania, United States